CLINICAL TRIAL: NCT00765076
Title: Observer-blind Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2186877A in Elderly Subjects
Brief Title: Clinical Study of the Immunogenicity of GSK Biologicals' Influenza Vaccine GSK2186877A in People Aged 65 Years or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112147
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Vaccine; Elderly; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- New generation influenza vaccine GSK2186877A Group (Experimental): Subjects aged ≥ 65 years receiving 1 dose of New generation influenza vaccine GSK2186877A at Day 0
  Interventions: Biological: GSK Biologicals' influenza vaccine GSK2186877A
- Fluarix elderly Group (Active Comparator): Subjects aged >= 65 years receiving 1 dose of Fluarix vaccine at Day 0
  Interventions: Biological: GSK Biologicals' Fluarix
- Fluarix young Group (Active Comparator): Subjects aged 18-40 years receiving 1 dose of Fluarix vaccine at Day 0
  Interventions: Biological: GSK Biologicals' Fluarix

INTERVENTIONS:
Biological: GSK Biologicals' influenza vaccine GSK2186877A — One intramuscular injection at Day 0
  Arms: New generation influenza vaccine GSK2186877A Group
Biological: GSK Biologicals' Fluarix — One intramuscular injection at Day 0
  Arms: Fluarix elderly Group; Fluarix young Group

SUMMARY:
This clinical trial aims to study the immunogenicity of GSK Biologicals' influenza vaccine GSK2186877A in people aged 65 years or older.

DETAILED DESCRIPTION:
The amendment to the protocol posting: minor change in one inclusion criterion and in one secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study. Specific attention should be given to the compliance potential of subjects with suspected or known drug or alcohol abuse.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by medical history and clinical examination before entering into the study.

Elderly adults:

• A man or woman 65 year of age or older at the time of the first vaccination.

Young adults:

* Man or woman between the ages of 18 and 40 years, inclusive.
* If the subject is female, she must be of non-childbearing potential or be post-menopausal, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to Visit 4 after vaccination and of an influenza vaccine other than the study vaccines up to Visit 4.
* Vaccination against influenza since February 2008 with a seasonal influenza vaccine.
* Previous vaccination in the last three years with an investigational adjuvanted vaccine candidate seasonal or pandemic influenza vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of hypersensivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s) including egg or chicken protein.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which intramuscular injections are contraindicated.
* Pregnant or lactating female.
* Female of childbearing age planning to become pregnant or planning to discontinue contraceptive precautions.
* Any medical condition that in the opinion of the investigator precludes the collection of blood volumes as required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-10-16; Primary Completion 2009-12-04 (Actual); Study Completion 2009-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Houston, Texas, United States
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Couch RB, Bayas JM, Caso C, Mbawuike IN, Lopez CN, Claeys C, El Idrissi M, Herve C, Laupeze B, Oostvogels L, Moris P. Superior antigen-specific CD4+ T-cell response with AS03-adjuvantation of a trivalent influenza vaccine in a randomised trial of adults aged 65 and older. BMC Infect Dis. 2014 Jul 30;14:425. doi: 10.1186/1471-2334-14-425. PMID 25078387
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Started | 69 | 73 | 50
Completed | 68 | 73 | 49
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 69 | 73 | 50 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (5.44) | 71.5 (5.32) | 26.0 (4.91) | 59.7 (20.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 27 | 92
  Male | 33 | 44 | 23 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean (GM) Number of Influenza-specific CD4 T-cells Per Million CD4+ T-cells Identified After in Vitro Stimulation With Pooled Vaccine Strains Which Are Producing at Least Two Different Markers
Description: The markers assessed were Cluster of Differentiation 40 Ligand (CD40L), interleukin-2 (IL-2), tumor necrosis factor alpha (TNF-α), interferon-gamma (IFN-γ)
Time Frame: Day 21
Population: Analysis was performed on According-to-Protocol (ATP) Immunogenicity cohort. This cohort included all evaluable subjects for whom data concerning immunogenicity were available. Analysis was only performed for New generation influenza vaccine GSK2186877A Group and Fluarix elderly Group.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4+ Tcells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 61 | 0
cells per million CD4+ Tcells | 3371.11 (3602.15) | 2108.10 (1728.38) |

2. Secondary Outcome: The GM Number of Influenza-specific CD4 T-cells Per Million CD4+ T-cells Identified After in Vitro Stimulation With Pooled Vaccine Strains and With Each Vaccine Strain Separately Which Were Producing at Least Two Different Markers
Description: The markers assessed were CD40L, IL-2, TNF-α, IFN-γ. The separate vaccine strains tested included A/Brisbane, A/Uruguay, B/Brisbane antigens.
Time Frame: At Day 0, 21, 42 and 180
Population: Analysis was performed on According-to-Protocol (ATP) Immunogenicity cohort. This cohort included all evaluable subjects for whom data concerning immunogenicity were available.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4+ Tcells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 64 | 44
cells per million CD4+ Tcells
  pooled vaccine strain Day 0: number analyzed (Participants) | 62 | 61 | 44
  pooled vaccine strain Day 0 | 1269.34 (1032.60) | 1309.30 (2098.97) | 2026.14 (1004.93)
  pooled vaccine strain Day 21: number analyzed (Participants) | 62 | 61 | 43
  pooled vaccine strain Day 21 | 3371.11 (3602.15) | 2108.10 (1728.38) | 3228.91 (1714.91)
  pooled vaccine strain Day 42: number analyzed (Participants) | 61 | 64 | 44
  pooled vaccine strain Day 42 | 2657.07 (1903.38) | 1540.08 (1138.94) | 2669.41 (1391.70)
  pooled vaccine strain Day 180: number analyzed (Participants) | 60 | 63 | 42
  pooled vaccine strain Day 180 | 2105.66 (1232.80) | 1484.11 (1024.53) | 2746.76 (1232.90)
  A/Brisbane vaccine strain Day 0: number analyzed (Participants) | 62 | 61 | 44
  A/Brisbane vaccine strain Day 0 | 402.28 (421.64) | 340.57 (352.55) | 793.58 (452.84)
  A/Brisbane vaccine strain Day 21: number analyzed (Participants) | 62 | 61 | 42
  A/Brisbane vaccine strain Day 21 | 1062.79 (1049.87) | 462.34 (712.32) | 982.18 (727.70)
  A/Brisbane vaccine strain Day 42: number analyzed (Participants) | 60 | 64 | 43
  A/Brisbane vaccine strain Day 42 | 822.07 (667.91) | 392.04 (498.81) | 874.34 (544.91)
  A/Brisbane vaccine strain Day 180: number analyzed (Participants) | 60 | 63 | 42
  A/Brisbane vaccine strain Day 180 | 669.67 (579.75) | 463.94 (458.04) | 973.29 (555.34)
  A/Uruguay vaccine strain Day 0: number analyzed (Participants) | 62 | 61 | 44
  A/Uruguay vaccine strain Day 0 | 342.58 (340.83) | 274.47 (282.29) | 437.07 (410.66)
  A/Uruguay vaccine strain Day 21: number analyzed (Participants) | 62 | 61 | 43
  A/Uruguay vaccine strain Day 21 | 930.98 (1262.81) | 497.49 (479.98) | 667.38 (465.08)
  A/Uruguay vaccine strain Day 42: number analyzed (Participants) | 59 | 64 | 44
  A/Uruguay vaccine strain Day 42 | 678.88 (669.99) | 331.62 (365.40) | 473.17 (500.92)
  A/Uruguay vaccine strain Day 180: number analyzed (Participants) | 59 | 62 | 41
  A/Uruguay vaccine strain Day 180 | 640.97 (567.70) | 331.02 (324.69) | 654.30 (503.69)
  B/Brisbane vaccine strain Day 0: number analyzed (Participants) | 61 | 61 | 44
  B/Brisbane vaccine strain Day 0 | 672.58 (615.67) | 504.36 (588.82) | 1183.48 (582.67)
  B/Brisbane vaccine strain Day 21: number analyzed (Participants) | 62 | 60 | 43
  B/Brisbane vaccine strain Day 21 | 1755.55 (1961.87) | 1149.98 (1032.36) | 1861.66 (884.81)
  B/Brisbane vaccine strain Day 42: number analyzed (Participants) | 58 | 62 | 44
  B/Brisbane vaccine strain Day 42 | 1325.35 (1094.01) | 807.46 (639.01) | 1572.47 (719.96)
  B/Brisbane vaccine strain Day 180: number analyzed (Participants) | 57 | 60 | 42
  B/Brisbane vaccine strain Day 180 | 1034.78 (725.84) | 778.13 (630.32) | 1640.71 (897.14)

3. Secondary Outcome: The GM Number of Influenza-specific CD4 T-cells Per Million CD4+ T-cells Identified After in Vitro Stimulation With Pooled Vaccine Strains and With Each Vaccine Strain Separately Producing Each of the Immune Markers Plus Another Immune Marker
Description: as for outcome 2
Time Frame: At Day 0, 21, 42 and 180
Population: The analysis was based on According-to-Protocol (ATP) Immunogenicity cohort which included all evaluable subjects for whom data concerning immunogenicity data were available.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4+ Tcells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 64 | 44
cells per million CD4+ Tcells
  pooled strain[CD4-CD40L] D 0: number analyzed (Participants) | 62 | 61 | 44
  pooled strain[CD4-CD40L] D 0 | 1104.24 (987.15) | 1211.72 (1086.88) | 1879.85 (963.74)
  pooled strain[CD4-CD40L] D 21: number analyzed (Participants) | 62 | 61 | 43
  pooled strain[CD4-CD40L] D 21 | 2817.50 (3166.07) | 1935.66 (1597.56) | 2929.86 (1644.61)
  pooled strain[CD4-CD40L] D 42: number analyzed (Participants) | 61 | 64 | 44
  pooled strain[CD4-CD40L] D 42 | 2447.37 (1766.85) | 1425.02 (1082.35) | 2436.43 (1365.81)
  pooled strain[CD4-CD40L] D 180: number analyzed (Participants) | 60 | 63 | 42
  pooled strain[CD4-CD40L] D 180 | 2036.70 (1170.14) | 1416.78 (973.63) | 2619.74 (1167.44)
  pooled strain[CD4- IFN-γ] D 0: number analyzed (Participants) | 62 | 61 | 44
  pooled strain[CD4- IFN-γ] D 0 | 832.47 (798.10) | 835.22 (1598.81) | 1403.57 (777.81)
  pooled strain[CD4- IFN-γ] D 21: number analyzed (Participants) | 62 | 61 | 43
  pooled strain[CD4- IFN-γ] D 21 | 2305.58 (2712.79) | 1341.17 (1195.01) | 2258.27 (1307.01)
  pooled strain[CD4- IFN-γ] D 42: number analyzed (Participants) | 61 | 64 | 44
  pooled strain[CD4- IFN-γ] D 42 | 1775.61 (1464.84) | 997.25 (818.08) | 1849.44 (1124.86)
  pooled strain[CD4- IFN-γ] D 180: number analyzed (Participants) | 60 | 63 | 42
  pooled strain[CD4- IFN-γ] D 180 | 1495.36 (1031.14) | 1019.64 (790.42) | 2102.93 (1074.53)
  pooled strain[CD4-IL-2] D 0: number analyzed (Participants) | 62 | 61 | 44
  pooled strain[CD4-IL-2] D 0 | 1085.32 (930.22) | 1119.34 (1002.46) | 1717.41 (852.57)
  pooled strain[CD4-IL-2] D 21: number analyzed (Participants) | 62 | 61 | 43
  pooled strain[CD4-IL-2] D 21 | 2534.86 (3188.65) | 1779.41 (1595.66) | 2690.36 (1583.12)
  pooled strain[CD4-IL-2] D42: number analyzed (Participants) | 61 | 64 | 44
  pooled strain[CD4-IL-2] D42 | 2205.91 (1754.74) | 1310.05 (1062.08) | 2199.18 (1251.48)
  pooled strain[CD4-IL-2] D 180: number analyzed (Participants) | 60 | 63 | 42
  pooled strain[CD4-IL-2] D 180 | 1837.60 (1093.26) | 1285.14 (955.76) | 2302.51 (1042.85)
  pooled strain[CD4-TNF-α] D 0: number analyzed (Participants) | 62 | 61 | 44
  pooled strain[CD4-TNF-α] D 0 | 874.43 (812.98) | 928.86 (1924.68) | 1425.50 (768.88)
  pooled strain[CD4-TNF-α] D 21: number analyzed (Participants) | 62 | 61 | 43
  pooled strain[CD4-TNF-α] D 21 | 2114.47 (2448.22) | 1284.20 (1080.26) | 1999.07 (1010.68)
  pooled strain[CD4-TNF-α] D 42: number analyzed (Participants) | 61 | 64 | 44
  pooled strain[CD4-TNF-α] D 42 | 1741.65 (1350.73) | 1012.42 (805.86) | 1752.99 (933.90)
  pooled strain[CD4-TNF-α] D 180: number analyzed (Participants) | 60 | 63 | 42
  pooled strain[CD4-TNF-α] D 180 | 1413.29 (865.27) | 1015.29 (830.38) | 1821.04 (880.59)
  A/Brisbane strain[CD4-CD40L] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Brisbane strain[CD4-CD40L] D 0 | 387.76 (400.63) | 320.29 (338.91) | 750.57 (435.67)
  A/Brisbane strain[CD4-CD40L] D 21: number analyzed (Participants) | 62 | 61 | 42
  A/Brisbane strain[CD4-CD40L] D 21 | 980.10 (937.63) | 462.64 (676.17) | 919.30 (679.26)
  A/Brisbane strain[CD4-CD40L] D 42: number analyzed (Participants) | 60 | 64 | 43
  A/Brisbane strain[CD4-CD40L] D 42 | 771.49 (616.20) | 365.94 (474.72) | 818.54 (522.72)
  A/Brisbane strain[CD4-CD40L] D 180: number analyzed (Participants) | 60 | 63 | 42
  A/Brisbane strain[CD4-CD40L] D 180 | 653.13 (547.36) | 466.55 (429.28) | 922.06 (511.19)
  A/Uruguay strain[CD4-CD40L] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Uruguay strain[CD4-CD40L] D 0 | 308.73 (316.94) | 227.76 (266.35) | 384.02 (397.54)
  A/Uruguay strain[CD4-CD40L] D 21: number analyzed (Participants) | 62 | 61 | 43
  A/Uruguay strain[CD4-CD40L] D 21 | 805.56 (1066.84) | 451.52 (459.24) | 602.51 (431.82)
  A/Uruguay strain[CD4-CD40L] D 42: number analyzed (Participants) | 59 | 64 | 44
  A/Uruguay strain[CD4-CD40L] D 42 | 592.88 (579.07) | 286.06 (333.05) | 417.15 (468.52)
  A/Uruguay strain[CD4-CD40L] D 180: number analyzed (Participants) | 59 | 62 | 41
  A/Uruguay strain[CD4-CD40L] D 180 | 609.34 (524.50) | 298.70 (295.58) | 584.68 (446.49)
  B/Brisbane strain[CD4-CD40L] D 0: number analyzed (Participants) | 61 | 61 | 44
  B/Brisbane strain[CD4-CD40L] D 0 | 647.94 (581.98) | 515.89 (566.11) | 1129.44 (573.40)
  B/Brisbane strain[CD4-CD40L] D 21: number analyzed (Participants) | 62 | 60 | 43
  B/Brisbane strain[CD4-CD40L] D 21 | 1607.98 (1806.43) | 1077.12 (990.77) | 1737.45 (842.62)
  B/Brisbane strain[CD4-CD40L] D 42: number analyzed (Participants) | 58 | 62 | 44
  B/Brisbane strain[CD4-CD40L] D 42 | 1246.10 (1033.85) | 763.04 (606.04) | 1472.48 (725.44)
  B/Brisbane strain[CD4-CD40L] D 180: number analyzed (Participants) | 57 | 60 | 42
  B/Brisbane strain[CD4-CD40L] D 180 | 1011.39 (682.07) | 757.17 (611.01) | 1570.98 (843.76)
  A/Brisbane strain[CD4- IFN-γ] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Brisbane strain[CD4- IFN-γ] D 0 | 279.24 (337.13) | 258.94 (258.55) | 563.26 (323.39)
  A/Brisbane strain[CD4- IFN-γ] D 21: number analyzed (Participants) | 62 | 61 | 42
  A/Brisbane strain[CD4- IFN-γ] D 21 | 725.55 (752.84) | 344.39 (447.19) | 680.40 (543.42)
  A/Brisbane strain[CD4- IFN-γ] D 42: number analyzed (Participants) | 60 | 64 | 43
  A/Brisbane strain[CD4- IFN-γ] D 42 | 572.87 (520.31) | 326.66 (322.73) | 623.21 (409.74)
  A/Brisbane strain[CD4- IFN-γ] D 180: number analyzed (Participants) | 60 | 63 | 42
  A/Brisbane strain[CD4- IFN-γ] D 180 | 586.26 (474.54) | 363.03 (361.43) | 773.40 (486.08)
  A/Uruguay strain[CD4- IFN-γ] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Uruguay strain[CD4- IFN-γ] D 0 | 214.92 (245.84) | 164.78 (199.00) | 283.81 (267.71)
  A/Uruguay strain[CD4- IFN-γ] D 21: number analyzed (Participants) | 62 | 61 | 43
  A/Uruguay strain[CD4- IFN-γ] D 21 | 641.94 (944.37) | 314.63 (311.72) | 403.00 (355.57)
  A/Uruguay strain[CD4- IFN-γ] D 42: number analyzed (Participants) | 59 | 64 | 44
  A/Uruguay strain[CD4- IFN-γ] D 42 | 458.72 (501.32) | 246.18 (227.80) | 331.47 (356.93)
  A/Uruguay strain[CD4- IFN-γ] D 180: number analyzed (Participants) | 59 | 62 | 41
  A/Uruguay strain[CD4- IFN-γ] D 180 | 426.59 (418.38) | 228.06 (215.33) | 451.90 (400.61)
  B/Brisbane strain[CD4- IFN-γ] D 0: number analyzed (Participants) | 61 | 61 | 44
  B/Brisbane strain[CD4- IFN-γ] D 0 | 342.59 (532.27) | 319.38 (507.10) | 824.76 (496.44)
  B/Brisbane strain[CD4- IFN-γ] D 21: number analyzed (Participants) | 62 | 60 | 43
  B/Brisbane strain[CD4- IFN-γ] D 21 | 1219.72 (1581.26) | 721.43 (849.49) | 1361.31 (712.84)
  B/Brisbane strain[CD4- IFN-γ] D 42: number analyzed (Participants) | 58 | 62 | 44
  B/Brisbane strain[CD4- IFN-γ] D 42 | 903.71 (918.49) | 517.83 (501.51) | 1095.12 (676.34)
  B/Brisbane strain[CD4- IFN-γ] D 180: number analyzed (Participants) | 57 | 60 | 42
  B/Brisbane strain[CD4- IFN-γ] D 180 | 697.03 (635.80) | 510.37 (539.79) | 1253.33 (862.51)
  A/Brisbane strain[CD4-IL2] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Brisbane strain[CD4-IL2] D 0 | 346.00 (369.76) | 319.16 (331.16) | 677.11 (397.23)
  A/Brisbane strain[CD4-IL2] D 21: number analyzed (Participants) | 62 | 61 | 42
  A/Brisbane strain[CD4-IL2] D 21 | 872.32 (897.70) | 427.26 (664.07) | 816.95 (655.93)
  A/Brisbane strain[CD4-IL2] D 42: number analyzed (Participants) | 60 | 64 | 43
  A/Brisbane strain[CD4-IL2] D 42 | 696.36 (598.29) | 393.67 (460.81) | 720.28 (468.43)
  A/Brisbane strain[CD4-IL2] D 180: number analyzed (Participants) | 60 | 63 | 42
  A/Brisbane strain[CD4-IL2] D 180 | 570.30 (503.83) | 387.63 (429.61) | 817.80 (470.25)
  A/Uruguay strain[CD4-IL2] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Uruguay strain[CD4-IL2] D 0 | 278.66 (306.46) | 240.26 (261.18) | 369.77 (322.49)
  A/Uruguay strain[CD4-IL2] D 21: number analyzed (Participants) | 62 | 61 | 43
  A/Uruguay strain[CD4-IL2] D 21 | 680.16 (1060.47) | 391.84 (425.96) | 510.88 (385.11)
  A/Uruguay strain[CD4-IL2] D 42: number analyzed (Participants) | 59 | 64 | 44
  A/Uruguay strain[CD4-IL2] D 42 | 534.07 (579.96) | 295.90 (322.75) | 438.09 (401.87)
  A/Uruguay strain[CD4-IL2] D 180: number analyzed (Participants) | 59 | 62 | 41
  A/Uruguay strain[CD4-IL2] D 180 | 526.12 (483.57) | 299.67 (274.20) | 514.55 (404.73)
  B/Brisbane strain[CD4-IL2] D 0: number analyzed (Participants) | 61 | 61 | 44
  B/Brisbane strain[CD4-IL2] D 0 | 587.16 (566.46) | 451.89 (549.60) | 1019.08 (512.69)
  B/Brisbane strain[CD4-IL2] D 21: number analyzed (Participants) | 62 | 60 | 43
  B/Brisbane strain[CD4-IL2] D 21 | 1496.41 (1826.01) | 1004.17 (966.20) | 1592.61 (810.35)
  B/Brisbane strain[CD4-IL2] D 42: number analyzed (Participants) | 58 | 62 | 44
  B/Brisbane strain[CD4-IL2] D 42 | 1144.72 (1021.68) | 724.10 (593.13) | 1322.64 (664.52)
  B/Brisbane strain[CD4-IL2] D 180: number analyzed (Participants) | 57 | 60 | 42
  B/Brisbane strain[CD4-IL2] D 180 | 933.06 (660.87) | 704.18 (602.50) | 1439.92 (753.90)
  A/Brisbane strain[CD4-TNF-α] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Brisbane strain[CD4-TNF-α] D 0 | 262.44 (349.53) | 247.22 (274.83) | 536.34 (369.21)
  A/Brisbane strain[CD4-TNF-α] D 21: number analyzed (Participants) | 62 | 61 | 42
  A/Brisbane strain[CD4-TNF-α] D 21 | 621.35 (746.04) | 289.38 (376.07) | 497.77 (499.72)
  A/Brisbane strain[CD4-TNF-α] D 42: number analyzed (Participants) | 60 | 64 | 43
  A/Brisbane strain[CD4-TNF-α] D 42 | 500.13 (518.12) | 238.28 (329.62) | 564.91 (395.51)
  A/Brisbane strain[CD4-TNF-α] D 180: number analyzed (Participants) | 60 | 63 | 42
  A/Brisbane strain[CD4-TNF-α] D 180 | 462.60 (402.23) | 308.96 (347.12) | 616.75 (383.70)
  A/Uruguay strain[CD4-TNF-α] D 0: number analyzed (Participants) | 62 | 61 | 44
  A/Uruguay strain[CD4-TNF-α] D 0 | 223.83 (292.61) | 191.52 (234.42) | 284.69 (317.94)
  A/Uruguay strain[CD4-TNF-α] D 21: number analyzed (Participants) | 62 | 61 | 43
  A/Uruguay strain[CD4-TNF-α] D 21 | 600.99 (932.13) | 320.59 (308.63) | 411.24 (333.50)
  A/Uruguay strain[CD4-TNF-α] D 42: number analyzed (Participants) | 59 | 64 | 44
  A/Uruguay strain[CD4-TNF-α] D 42 | 452.35 (515.50) | 211.12 (267.39) | 333.52 (375.97)
  A/Uruguay strain[CD4-TNF-α] D 180: number analyzed (Participants) | 59 | 62 | 41
  A/Uruguay strain[CD4-TNF-α] D 180 | 370.86 (415.54) | 230.70 (241.03) | 477.18 (355.92)
  B/Brisbane strain[CD4-TNF-α] D 0: number analyzed (Participants) | 61 | 61 | 44
  B/Brisbane strain[CD4-TNF-α] D 0 | 414.10 (472.20) | 305.51 (516.15) | 773.44 (420.89)
  B/Brisbane strain[CD4-TNF-α] D 21: number analyzed (Participants) | 62 | 60 | 43
  B/Brisbane strain[CD4-TNF-α] D 21 | 967.79 (1226.62) | 639.74 (663.66) | 1057.83 (507.15)
  B/Brisbane strain[CD4-TNF-α] D 42: number analyzed (Participants) | 58 | 62 | 44
  B/Brisbane strain[CD4-TNF-α] D 42 | 775.92 (756.63) | 413.38 (490.41) | 953.30 (491.50)
  B/Brisbane strain[CD4-TNF-α] D 180: number analyzed (Participants) | 57 | 60 | 42
  B/Brisbane strain[CD4-TNF-α] D 180 | 642.05 (520.83) | 475.44 (511.57) | 1051.51 (664.61)

4. Secondary Outcome: Haemagglutinin Inhibition (HI) Antibody Titers
Description: Antibody titers were expressed as Geometric mean titers (GMTs) calculated after invitro stimulation with separate vaccine strains.
Time Frame: At Day 0, 21, 42 and 180
Population: The analysis of immunogenicity was performed on According-to-Protocol (ATP) Immunogenicity cohort which included all evaluable subjects for whom data concerning immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 66 | 44
titer
  A/Brisbane strain at Day 0 | 16.5 [12.7 to 21.5] | 14.3 [10.9 to 18.7] | 20.5 [13.0 to 32.3]
  A/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 21 | 105.1 [80.3 to 137.6] | 67.2 [49.6 to 91.2] | 220.8 [163.3 to 298.7]
  A/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Brisbane strain at Day 42 | 82.3 [64.5 to 105.0] | 56.8 [42.0 to 77.0] | 181.4 [133.5 to 246.6]
  A/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 180 | 38.4 [30.3 to 48.7] | 32.1 [24.0 to 42.8] | 90.3 [60.7 to 134.2]
  A/Uruguay strain at Day 0 | 21.4 [15.0 to 30.4] | 17.5 [13.2 to 23.3] | 16.4 [11.0 to 24.5]
  A/Uruguay strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 21 | 330.9 [239.8 to 456.7] | 164.2 [113.3 to 238.0] | 179.0 [115.1 to 278.4]
  A/Uruguay strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Uruguay strain at Day 42 | 254.8 [182.1 to 356.5] | 110.1 [77.4 to 156.6] | 130.3 [86.6 to 196.1]
  A/Uruguay strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 180 | 117.0 [83.0 to 164.9] | 59.9 [41.8 to 85.9] | 74.4 [47.6 to 116.2]
  B/Brisbane strain at Day 0 | 92.0 [66.2 to 127.8] | 97.0 [72.9 to 129.2] | 169.0 [108.2 to 263.9]
  B/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 21 | 699.9 [538.4 to 909.8] | 502.6 [388.6 to 650.0] | 1229.4 [972.8 to 1553.8]
  B/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  B/Brisbane strain at Day 42 | 487.2 [372.2 to 637.8] | 393.9 [310.3 to 500] | 971.6 [778.0 to 1213.3]
  B/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 180 | 254.5 [195.3 to 331.6] | 238.4 [188.4 to 301.6] | 677.2 [513.7 to 892.7]

5. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies Calculated After in Vitro Stimulation With Separate Vaccine Strains.
Description: Seropositivity was defined as antibody titer greater than or equal to the cut-off value i.e ≥ 1:10
Time Frame: At Day 0, 21, 42 and 180
Population: The analysis was performed on According-to-Protocol (ATP) immunogenicity cohort which included all evaluable subjects for whom data concerning immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 66 | 44
Participants
  A/Brisbane strain at Day 0 | 43 | 40 | 25
  A/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 21 | 61 | 62 | 43
  A/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Brisbane strain at Day 42 | 60 | 62 | 44
  A/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 180 | 57 | 57 | 40
  A/Uruguay strain at Day 0 | 41 | 45 | 24
  A/Uruguay strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 21 | 62 | 63 | 41
  A/Uruguay strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Uruguay strain at Day 42 | 60 | 62 | 42
  A/Uruguay strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 180 | 61 | 59 | 39
  B/Brisbane strain at Day 0 | 59 | 65 | 42
  B/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 21 | 62 | 66 | 43
  B/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  B/Brisbane strain at Day 42 | 61 | 65 | 44
  B/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 180 | 62 | 66 | 43

6. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies
Description: Seroconversion was defined as the number of vaccinees who had either a prevaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 21, 42 and 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 66 | 44
Participants
  A/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 21 | 36 | 32 | 29
  A/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Brisbane strain at Day 42 | 33 | 25 | 29
  A/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 180 | 16 | 16 | 23
  A/Uruguay strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 21 | 52 | 50 | 33
  A/Uruguay strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Uruguay strain at Day 42 | 48 | 44 | 30
  A/Uruguay strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 180 | 36 | 28 | 20
  B/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 21 | 44 | 38 | 29
  B/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  B/Brisbane strain at Day 42 | 38 | 35 | 25
  B/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 180 | 22 | 22 | 20

7. Secondary Outcome: HI Antibody Seroconversion Factors
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0.
Time Frame: At Day 21, 42 and 180
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 66 | 44
fold increase
  A/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 21 | 6.4 [4.5 to 9.0] | 4.7 [3.4 to 6.6] | 10.6 [6.3 to 17.9]
  A/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Brisbane strain at Day 42 | 5.1 [3.7 to 7.0] | 3.9 [2.8 to 5.4] | 8.9 [5.3 to 14.7]
  A/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 180 | 2.3 [1.8 to 3.0] | 2.2 [1.7 to 3.0] | 4.6 [2.9 to 7.2]
  A/Uruguay strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 21 | 15.5 [10.8 to 22.2] | 9.4 [6.6 to 13.2] | 11.3 [7.2 to 17.8]
  A/Uruguay strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Uruguay strain at Day 42 | 12.2 [8.5 to 17.4] | 6.4 [4.7 to 8.6] | 7.9 [5.3 to 11.9]
  A/Uruguay strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 180 | 5.5 [4.1 to 7.3] | 3.4 [2.5 to 4.6] | 4.5 [3.0 to 6.9]
  B/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 21 | 7.6 [5.6 to 10.3] | 5.2 [3.8 to 7.1] | 7.4 [4.7 to 11.6]
  B/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  B/Brisbane strain at Day 42 | 5.4 [4.0 to 7.2] | 4.1 [3.1 to 5.4] | 5.8 [3.7 to 8.9]
  B/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 180 | 2.8 [2.2 to 3.4] | 2.5 [1.9 to 3.1] | 4.0 [2.8 to 5.8]

8. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: At Day 0, 21, 42 and 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 62 | 66 | 44
Participants
  A/Brisbane strain at Day 0 | 20 | 16 | 18
  A/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 21 | 57 | 53 | 42
  A/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Brisbane strain at Day 42 | 56 | 47 | 42
  A/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Brisbane strain at Day 180 | 39 | 34 | 36
  A/Uruguay strain at Day 0 | 26 | 24 | 16
  A/Uruguay strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 21 | 61 | 57 | 39
  A/Uruguay strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  A/Uruguay strain at Day 42 | 59 | 53 | 39
  A/Uruguay strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  A/Uruguay strain at Day 180 | 53 | 48 | 33
  B/Brisbane strain at Day 0 | 51 | 57 | 39
  B/Brisbane strain at Day 21: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 21 | 62 | 65 | 43
  B/Brisbane strain at Day 42: number analyzed (Participants) | 61 | 65 | 44
  B/Brisbane strain at Day 42 | 61 | 64 | 44
  B/Brisbane strain at Day 180: number analyzed (Participants) | 62 | 66 | 43
  B/Brisbane strain at Day 180 | 60 | 65 | 42

9. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling was >100mm and grade 3 pain was considerable pain at rest, that prevented normal everyday activity.
Time Frame: Day 0 -6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants
  Any ecchymosis | 2 | 1 | 0
  Grade 3 ecchymosis | 0 | 0 | 0
  Any pain | 43 | 15 | 35
  Grade 3 pain | 0 | 0 | 0
  Any redness | 5 | 0 | 0
  Grade 3 redness | 0 | 0 | 0
  Any swelling | 8 | 1 | 0
  Grade 3 swelling | 0 | 0 | 0

10. Secondary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as the number of days with any grade of local symptoms.
Time Frame: Day 0 -6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented on subjects who experienced the symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 43 | 15 | 35
Days
  Ecchymosis: number analyzed (Participants) | 2 | 1 | 0
  Ecchymosis | 3.5 [3.0 to 4.0] | 5.0 [5.0 to 5.0] |
  Pain | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Redness: number analyzed (Participants) | 5 | 0 | 0
  Redness | 2.0 [1.0 to 5.0] |  |
  Swelling: number analyzed (Participants) | 8 | 1 | 0
  Swelling | 4.0 [1.0 to 6.0] | 5.0 [5.0 to 5.0] |

11. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any fever was defined as oral temperature ≥ 38.0 degree centigrade (°C), grade 3 fever was defined as oral temperature ≥ 39.0°C. For other symptoms grade 3 was defined as general symptom that prevented normal activity and related was general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0 -6
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants
  Any arthralgia | 14 | 3 | 4
  Grade 3 arthralgia | 0 | 0 | 0
  Related arthralgia | 12 | 1 | 3
  Any fatigue | 22 | 12 | 21
  Grade 3 fatigue | 0 | 0 | 0
  Related fatigue | 21 | 8 | 11
  Any gastrointestinal symptoms | 6 | 4 | 6
  Grade 3 gastrointestinal symptoms | 0 | 0 | 0
  Related gastrointestinal symptoms | 5 | 1 | 4
  Any headache | 22 | 7 | 14
  Grade 3 headache | 0 | 0 | 0
  Related headache | 17 | 2 | 7
  Any myalgia | 17 | 8 | 11
  Grade 3 myalgia | 0 | 0 | 0
  Related myalgia | 16 | 7 | 9
  Any shivering | 11 | 0 | 2
  Grade 3 shivering | 0 | 0 | 1
  Related shivering | 8 | 0 | 1
  Any fever | 2 | 0 | 0
  Grade 3 fever | 1 | 0 | 0
  Related fever | 2 | 0 | 0

12. Secondary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: Day 0 -6
Population: as for outcome 10
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 22 | 12 | 21
Days
  Arthralgia: number analyzed (Participants) | 14 | 3 | 4
  Arthralgia | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 6.0]
  Fatigue | 2.0 [1.0 to 7.0] | 2.5 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 6 | 4 | 6
  Gastrointestinal symptoms | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Headache: number analyzed (Participants) | 22 | 7 | 14
  Headache | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 4.0] | 1.5 [1.0 to 4.0]
  Myalgia: number analyzed (Participants) | 17 | 8 | 11
  Myalgia | 2.0 [1.0 to 6.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Shivering: number analyzed (Participants) | 11 | 0 | 2
  Shivering | 1.0 [1.0 to 7.0] |  | 2.5 [2.0 to 3.0]
  Fever: number analyzed (Participants) | 2 | 0 | 0
  Fever | 2.0 [1.0 to 3.0] |  |

13. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom, regardless of intensity or relation to vaccination, grade 3 was unsolicited symptom that prevented normal activity and related was event assessed by investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants
  Any AE(s) | 13 | 21 | 15
  Grade 3 AE(s) | 2 | 2 | 1
  Related AE(s) | 3 | 2 | 1

14. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit (MAEs)
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom, regardless of intensity or relation to vaccination, grade 3 was defined as symptom that prevented normal activity and related was event assessed by investigator as causally related to the study vaccination.
Time Frame: Day 0-179
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants
  Any MAE(s) | 24 | 21 | 13
  Grade 3 MAE(s) | 4 | 9 | 3
  Related MAE(s) | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects Reporting Any AEs of Specific Interest (AESI)
Description: AESI for safety monitoring are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Any was defined as occurrence of any symptom, regardless of intensity or relation to vaccination.
Time Frame: Day 0-364
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom, regardless of intensity or relation to vaccination and related was event assessed by investigator as causally related to the study vaccination.
Time Frame: Day 0-364
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 69 | 73 | 50
Participants | 5 | 11 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to day 364. Systematically assessed frequent adverse events (AEs) were assessed during 7 day post vaccination period. Non systematically assessed frequent AEs were assessed during 21 day post vaccination period.
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 5/69 | 11/73 | 1/50
Other Adverse Events (participants affected / at risk) | 53/69 | 27/73 | 43/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=69) | Fluarix Elderly Group (N=73) | Fluarix Young Group (N=50)
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=69) | Fluarix Elderly Group (N=73) | Fluarix Young Group (N=50)
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4
Pain (General disorders) | 43 | 15 | 35
Redness (General disorders) | 5 | 0 | 0
Swelling (General disorders) | 8 | 1 | 0
Arthralgia (General disorders) | 14 | 3 | 4
Fatigue (General disorders) | 22 | 12 | 21
Gastrointestinal symptoms (General disorders) | 6 | 4 | 6
Headache (General disorders) | 22 | 7 | 14
Myalgia (General disorders) | 17 | 8 | 11
Shivering (General disorders) | 11 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.